CLINICAL TRIAL: NCT00852202
Title: A Double-blind, Placebo-controlled Study of RGH-188 (Cariprazine) in Bipolar Depression
Brief Title: Safety and Efficacy of RGH-188 (Cariprazine) in Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-52
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Depression
Keywords: bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 0.25 - 0.75 mg/day cariprazine capsules, oral administration, once daily dosing.
  Interventions: Drug: cariprazine
- 2 (Experimental): 1.5 - 3.0 mg/day cariprazine capsules, oral administration, once daily dosing.
  Interventions: Drug: cariprazine
- 3 (Placebo Comparator): Matching placebo capsules, oral administration, once daily dosing.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cariprazine — Drug: cariprazine (0.25 - 0.75 mg/day)
  Arms: 1
Drug: cariprazine — Drug: cariprazine (1.5 - 3.0 mg/day)
  Arms: 2
Drug: placebo — placebo capsules, oral administration, once daily dosing
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of cariprazine in the treatment of outpatients with bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old
* Currently meet the DSM-IV-TR criteria for Bipolar I or II Disorder without psychotic features, with a current depressive episode
* A verified previous manic, hypomanic, or mixed episode
* Score of 20 or higher on the HAMD-17
* Score of 2 or higher on Item 1 of the HAMD

Exclusion Criteria:

* Score greater than 12 on the Young Mania Rating Scale
* Eight or more episodes of a mood disturbance (depression, mania, hypomania, or mixed state) within the 12 months prior to Visit 1
* Principal DSM-IV-TR-based diagnosis of an axis I disorder other than bipolar disorder (a secondary diagnosis of comorbid Generalized Anxiety Disorder, Social Anxiety Disorder, or specific phobias is acceptable)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2010-06-15 (Actual); Study Completion 2010-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Greenberg, MD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (26):
- United States (26):
  - Forest Investigative Site 005, Encino, California
  - Forest Investigative Site 017, Garden Grove, California
  - Forest Investigative Site 027, National City, California
  - Forest Investigative Site 013, Newport Beach, California
  - Forest Investigative Site 010, Oceanside, California
  - Forest Investigative Site 020, Bradenton, Florida
  - Forest Investigative Site 007, Jacksonville, Florida
  - Forest Investigative Site 019, Kissimmee, Florida
  - Forest Investigative Site 026, Orlando, Florida
  - Forest Investigative Site 012, West Palm Beach, Florida
  - Forest Investigative Site 024, Glen Burnie, Maryland
  - Forest Investigative Site 029, Creve Coeur, Missouri
  - Forest Investigative Site 002, Omaha, Nebraska
  - Forest Investigative Site 028, Cherry Hill, New Jersey
  - Forest Investigative Site 001, The Bronx, New York
  - Forest Investigative Site 018, Durham, North Carolina
  - Forest Investigative Site 004, Dayton, Ohio
  - Forest Investigative Site 022, Mason, Ohio
  - Forest Investigative Site 015, Portland, Oregon
  - Forest Investigative Site 006, Media, Pennsylvania
  - Forest Investigative Site 011, Philadelphia, Pennsylvania
  - Forest Investigative Site 014, Nashville, Tennessee
  - Forest Investigative Site 023, Irving, Texas
  - Forest Investigative Site 003, Woodstock, Vermont
  - Forest Investigative Site 009, Bellevue, Washington
  - Forest Investigative Site 016, Seattle, Washington

REFERENCES:
- [Derived] Earley WR, Burgess M, Rekeda L, Hankinson A, McIntyre RS, Suppes T, Calabrese JR, Yatham LN. A pooled post hoc analysis evaluating the safety and tolerability of cariprazine in bipolar depression. J Affect Disord. 2020 Feb 15;263:386-395. doi: 10.1016/j.jad.2019.11.098. Epub 2019 Nov 22. PMID 31969269

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 233 patients were randomized to receive double-blind treatment, 227 patients received at least 1 dose of double-blind treatment and were included in safety Population
Groups:
- Placebo: Matching placebo capsules, orally administered for 8 weeks
- 0.25 to 0.75 mg Cariprazine: Cariprazine capsules 0.25 to 0.75 mg was orally administrated once daily for 8 weeks
- 1.5 to 3.0 mg Cariprazine: 1.5 to 3.0 mg Cariprazine capsules, orally administrated once daily for 8 weeks
Period: Overall Study
Arm/Group | Placebo | 0.25 to 0.75 mg Cariprazine | 1.5 to 3.0 mg Cariprazine
Started | 77 | 75 | 75
Completed | 60 | 63 | 49
Not Completed | 17 | 12 | 26
Not completed — Adverse Event | 2 | 3 | 7
Not completed — Lack of Efficacy | 4 | 1 | 2
Not completed — Protocol Violation | 2 | 2 | 7
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Lost to Follow-up | 5 | 5 | 6
Not completed — pregnancy,moving away and surgery | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 1.5 to 3.0 mg Cariprazine: Cariprazine capsules 1.5 to 3.0 mg was orally administrated once daily for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.25 to 0.75 mg Cariprazine | 1.5 to 3.0 mg Cariprazine | Total
Number analyzed (Participants) | 77 | 75 | 75 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (10.7) | 37.4 (10.7) | 38.8 (12.1) | 38.9 (11.2)
Age, Customized [Number; unit: Participants]
  < 20 | 1 | 1 | 2 | 4
  20, 30 | 11 | 21 | 18 | 50
  30, 40 | 24 | 20 | 20 | 64
  40, 50 | 23 | 23 | 20 | 66
  50, 60 | 17 | 10 | 13 | 40
  ≥ 60 | 1 | 0 | 2 | 3
Sex/Gender, Customized [Number; unit: participant]
  Female | 46 | 48 | 51 | 145
  Male | 31 | 27 | 24 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 6 | 13
  Not Hispanic or Latino | 74 | 71 | 69 | 214
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 54 | 56 | 62 | 172
  Non-Caucasian | 23 | 19 | 13 | 55
  Black | 19 | 16 | 11 | 46
  Asian | 2 | 2 | 1 | 5
  Other | 2 | 1 | 1 | 4
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The patient is rated on a scale from 0-6 on 10 items. Apparent sadness, reported sadness, lassitude, pessimistic thoughts, inner tension, suicidal thoughts, reduced sleep and appetite, concentration difficulties, inability to feel. The overall MADRS score ranges from 0-60, with 0 meaning no symptoms and score of 60 meaning maximum severity.
Time Frame: Baseline to Week 8
Population: of the 227 included to the safety population, the mixed-effects model for repeated measures (MMRM) of the Intent to Treat study population was 60 for placebo, 64 for 0.25-0.75 mg Cariprazine and 54 for 1.5 to 3.0 mg Cariprazine
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | 0.25 to 0.75 mg Cariprazine | 1.5 to 3.0 mg Cariprazine
Number analyzed (Participants) | 60 | 64 | 54
Score on scale | 29.9 (0.6) | 30.2 (0.6) | 30.9 (0.6)
Statistical Analysis 1: Comparison: Placebo vs 0.25 to 0.75 mg Cariprazine; Test type: Superiority; p = 0.7408, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 1.5 to 3.0 mg Cariprazine; Test type: Superiority; p = 0.9961, ANCOVA

2. Secondary Outcome: Change in Baseline in Clinical Global Impressions-Improvement ( CGI-I )
Description: The patient was rated on a scale from 1 to 7, with 1 indicating the patient was very much improved and 7 indicating that the patient was very much worse.
Time Frame: Baseline to Week 8
Population: of the 227 included to the safety population, the mixed-effects model for repeated measures (MMRM) of the Intent to Treat study population was 60 for placebo, 64 for 0.25-0.75 mg Cariprazine and 53 for 1.5 to 3.0 mg Cariprazine
Measure: Mean (Standard Error); unit: Score on Scale
Groups:
- 1.5 to 3.0mg Cariprazine: Cariprazine capsules 1.5 to 3.0 mg was orally administrated once daily for 8 weeks
Arm/Group | Placebo | 0.25 to 0.75 mg Cariprazine | 1.5 to 3.0mg Cariprazine
Number analyzed (Participants) | 60 | 64 | 74
Score on Scale | 2.1 (0.1) | 2.1 (0.1) | 2.1 (0.2)
Statistical Analysis 1: Comparison: Placebo vs 0.25 to 0.75 mg Cariprazine; Test type: Superiority; p = 0.3441, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 1.5 to 3.0mg Cariprazine; Test type: Superiority; p = 0.2683, ANCOVA

ADVERSE EVENTS:
Arm/Group | Placebo | 0.25 to 0.75 mg Cariprazine | 1.5 to 3.0 mg Cariprazine
Serious Adverse Events (participants affected / at risk) | 2/77 | 2/75 | 2/75
Other Adverse Events (participants affected / at risk) | 51/77 | 48/75 | 52/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | 0.25 to 0.75 mg Cariprazine (N=75) | 1.5 to 3.0 mg Cariprazine (N=75)
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Suicidal attempt (Psychiatric disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | 0.25 to 0.75 mg Cariprazine (N=75) | 1.5 to 3.0 mg Cariprazine (N=75)
Insomnia (Psychiatric disorders) | 7 | 13 | 15
Akathisia (Nervous system disorders) | 5 | 2 | 13
Headache (Nervous system disorders) | 12 | 11 | 12
Nausea (Gastrointestinal disorders) | 4 | 9 | 9
Nasopharyngitis (Infections and infestations) | 5 | 7 | 7
Fatigue (General disorders) | 5 | 7 | 6
Weight Increase (Investigations) | 1 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 5
Anxiety (Psychiatric disorders) | 5 | 2 | 5
Restlessness (Psychiatric disorders) | 3 | 2 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Dry mouth (Gastrointestinal disorders) | 4 | 7 | 10
Migraine (Nervous system disorders) | 1 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 11 | 8
Constipation (Gastrointestinal disorders) | 5 | 5 | 3
Flatulence (Gastrointestinal disorders) | 4 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 2 | 3
Dysgeusia (Nervous system disorders) | 4 | 1 | 2
Sedation (Nervous system disorders) | 5 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.